CLINICAL TRIAL: NCT00442988
Title: Early Prediction of New Onset Diabetes Mellitus After Transplantation (NODAT) in Renal Transplantation: Use of Oral Glucose Tolerance Test (OGTT) and Fasting Plasma Glucose (FPG).
Brief Title: Prediction of NODAT After Renal Transplantation
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Other Study IDs: NODAT
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2007-03

CONDITIONS: Renal Transplantation
Keywords: NODAT; OGTT; FPG; Renal Transplanation; Risk Factors; Predictive value

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A statistical analysis of the predictive value of OGTT and FPG testing executed as part of standard clinical practice after renal transplantation for the diagosis of new-onset diabetes mellitus after transplantation.

DETAILED DESCRIPTION:
All patients transplanted in our department receive a formal oral glucose tolerance test (and thus also fasting plasma glucose concentration) in the first week after renal transplantation. This testing for DM or Impaired Glucose Tolerance (IGT) is part of our standard clinical protocol and data are collected prospectively in all these patients in an electronic patient medical file. The development of diabetes mellitus in all transplant patients is documented, including DM therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary single kidney transplantation
* Age older than 18 years

Exclusion Criteria:

* Pre-existing DM or documented impaired glucose metabolism
* Combined organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2000-10; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Dirk R Kuypers, MD, PhD, Principal Investigator — Department of Nephrology and Renal Transplantation, University Hospitals Leuven, Belgium
Locations (1):
- Dpt of Nephrology and Renal Transplantation, Leuven, Belgium